CLINICAL TRIAL: NCT00109733
Title: A Phase IIIb, Prospective, Multicenter, Randomized, Open-label Study to Determine the Safety and Efficacy of Two Different Dosing Regimens of Saizen® (Recombinant Human Growth Hormone (r-hGH), Using Cool.Click™ in Subjects With Childhood-onset Growth Hormone Deficiency During the Adolescent Transition Phase (CATS)
Brief Title: Cool.Click™ Adolescent Transition Study: Study of Saizen® in Subjects With Childhood-onset Growth Hormone Deficiency
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: EMD Serono (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 25253
Record Dates: First submitted 2005-05-02; First posted 2005-05-03 (Estimated); Results first posted 2010-06-22 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2013-08

CONDITIONS: Childhood-onset Growth Hormone Deficiency; Pituitary Dwarfism
Keywords: Childhood-onset growth hormone deficiency (COGHD); Saizen®
MeSH Terms: conditions — Dwarfism, Pituitary | interventions — Growth Hormone; Human Growth Hormone

ARMS (2):
- Standard dose group (Experimental): 0.005 mg/kg/day recombinant human growth hormone (r-hGH) for 30 days then increasing, with the Investigator's approval, to 0.010 mg/kg/day from Day 31 to Week 24.
  Interventions: Biological: recombinant human growth hormone
- High dose group (Experimental): 0.010 mg/kg/day recombinant human growth hormone for 14 days with the opportunity to dose escalate, with the Investigator's approval, on Day 15 to 0.02 mg/kg/day and Day 29 to 0.03 mg/kg/day.
  Interventions: Biological: recombinant human growth hormone

INTERVENTIONS:
Biological: recombinant human growth hormone — 0.005 mg/kg/day for 30 days then increasing, with the Investigator's approval, to 0.010 mg/kg/day from Day 31 to Week 24.
  Other Names: Saizen; r-hGH; cool click
  Arms: Standard dose group
Biological: recombinant human growth hormone — 0.010 mg/kg/day for 14 days with the opportunity to dose escalate, with the Investigator's approval, on Day 15 to 0.02 mg/kg/day and Day 29 to 0.03 mg/kg/day.
  Other Names: Saizen; r-hGH; cool click
  Arms: High dose group

SUMMARY:
The primary objective is to evaluate the efficacy and safety of two different dose regimens of r-hGH (Saizen®) in subjects with childhood-onset growth hormone deficiency (COGHD) during the transition phase from childhood to adulthood.

DETAILED DESCRIPTION:
This is a phase IIIb, prospective, multicenter, randomised, open label study to determine the safety and efficacy of two different dose regimens of r-hGH with a dose escalation scheme. Screening assessments must be completed 30 days prior to SD1 (Study Day 1). Eligible subjects ages 13 to 25 years will be randomised in equal allocation in a 1:1 ratio to one of two treatment groups (30 subjects/group). Daily subcutaneous injections will be self-administered or received from a designated individual using cool.click™, the needle-free growth hormone (GH) delivery device. The study consists of three periods: screening (up to 30 days prior to Study Day 1), active treatment (up to 24 weeks), and follow-up (4 week safety evaluation after the last dose of study medication).

Each subject will be required to complete a daily treatment diary to assess dosing compliance, adverse events, and concomitant medications. Each subject will receive one treatment diary at SD1, weeks 8, 12, and 24. Subjects will be required to record daily diary entries that will capture dosing compliance, adverse events, and concomitant medications. Depending upon treatment allocation and subject tolerability, dose titration will be increased as follows:

* Group A: 0.005 mg/kg/day for 30 days then increasing, with the Investigator's approval, to 0.010 mg/kg/day from day 31 to week 24.
* Group B: 0.010 mg/kg/day for 14 days with the opportunity to dose escalate, with the Investigator's approval, on day 15 to 0.02 mg/kg/day and day 29 to 0.03 mg/kg/day.

Scheduled study visits include screening, baseline, and weeks 8, 12, and 24. Dosage adjustments will be based on subject tolerability and telephone assessments from study drug initiation through week 6. Trunk fat will be measured at SD1, weeks 12 and 24 (or early termination visit). Routine clinical laboratory assessments (hematology, blood chemistries, and urinalysis) will be performed pre-treatment (-30 to -1 SD1) and post-treatment on week 24 (or early termination visit). Special laboratory assessments include the central analysis of lipid panel, fasting insulin, fasting glucose, insulin-like growth factor I (IGF-I), insulin-like growth factor binding protein 3 (IGFBP-3), free thyroxine (T4) , total T4, C-reactive protein (CRP). Physical exams will be performed at screening, weeks 12 and 24. Safety evaluations will occur during scheduled study visits, through telephone assessments, and by the review of adverse events and concomitant events on the subject treatment diary.

ELIGIBILITY:
Inclusion Criteria:

The day of entry or Study Day 1 is defined as the first day of study treatment. To be eligible for inclusion into this study, the subjects must fulfill all of the following criteria within 30 days prior to Study Day 1.

* Male or female from 13 to 25 years of age, inclusive
* Diagnosis of childhood onset growth hormone deficiency (GHD) and prior completed growth hormone (GH) treatment as evidenced by bone age greater than 14 years for girls and 16 years for boys or no height increase > 0.5 cm in the 6 months prior to Screen.
* Have documented GH deficiency (acquired or idiopathic), established by a standard provocative test, such as insulin (<5 ng/mL) or growth hormone releasing hormone plus arginine (<9 ng/mL) at least 30 days after GH has been discontinued. If a subject is hypopituitary with two or more pituitary disorders and has a low IGF-1, the stimulation test does not need to be performed to confirm GHD.
* If hypopituitary, must have been on adequate replacement therapy (if required) of glucocorticosteroids, thyroid and sex hormones (hormone levels on replacement being in normal/mildly elevated range) for at least 6 months prior to Screen.
* Be willing and able to comply with the protocol for the duration of the study.
* Have given written informed consent before any study-related procedure not part of the subject's normal medical care, with the understanding that the subject may withdraw consent at any time without prejudice to future medical care.
* Female subjects of childbearing potential must use a hormonal contraceptive, intra-uterine device, diaphragm with spermicide or condom with spermicide for the duration of the study. Confirmation that a female patient is not pregnant must be established by a negative human chorionic gonadotrophin (hCG) pregnancy test (urine or serum) within 7 days of study enrolment (SD1).

Exclusion Criteria:

To be eligible for inclusion in this study the subjects must not meet any of the following criteria:

* Known allergy or hypersensitivity to growth hormone or diluent.
* Previous treatment with GH within six months prior to Screen.
* Severe illness during the previous six months.
* Active malignancy (except non-melanomatous skin malignancies).
* Diabetes mellitus (type I or II).
* Seropositivity for human immunodeficiency virus (HIV), Hepatitis B surface antigen (HbsAg) and/or Hepatitis C Virus (HCV) serology.
* Pregnancy or lactation.
* History of drug and/or alcohol abuse or use of drugs for non-therapeutic purposes.
* Any medical condition that, in the opinion of the Investigator, would jeopardize the patient's safety following exposure to study drug.
* Clinically significant abnormal hematology, chemistry or urinalysis results at screening in the judgment of the Investigator.
* Have taken another investigational drug or had any experimental procedure in the six months preceding study entry.

Ages: 13 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 31 (Actual)
Dates: Start 2005-01; Primary Completion 2006-06 (Actual); Study Completion 2006-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sanja Dragnic, MD, Study Director — EMD Serono
Locations (9):
- United States (9):
  - Children's Hospital of Orange County, Orange, California
  - Nemours Children's Clinic, Jacksonville, Florida
  - Nemours Children's Clinic, Orlando, Florida
  - Pediatric Endocrinology Children's Clinic, Tallahassee, Florida
  - Pediatric Endocrine Associates, Atlanta, Georgia
  - Women's and Children's Hospital of Buffalo, Buffalo, New York
  - Columbia University, New York, New York
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- See also: Full FDA approved prescribing information can be found here — http://www.saizenus.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study Initiation Date: 06 Jan 2005 (date of first subject, first dose) Study Completion Date 11 Jun 2006 (date of last subject, last visit) 19 study centres in the United States received IRB approval to participate in this study; 13 of the centres enrolled at least one subject into the study.
Pre-assignment Details: All study screening assessments were to be performed within a 30-day period prior to study entry. A total of 40 subjects were screened for the study and 31 of them (77.5%) were randomised and received study drug.
Groups:
- Standard Dose Group: 0.005 mg/kg/day recombinant human growth hormone(r-hGH)for 30 days then increasing, with the Investigator's approval, to 0.010 mg/kg/day from Day 31 to Week 24.
Period: Overall Study
Arm/Group | Standard Dose Group | High Dose Group
Started | 15 | 16
Completed | 13 | 12
Not Completed | 2 | 4
Not completed — Protocol Violation | 0 | 1
Not completed — Stopped taking study drug | 1 | 1
Not completed — Non-compliant | 0 | 1
Not completed — Could not commit time for study | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Dose Group | High Dose Group | Total
Number analyzed (Participants) | 15 | 16 | 31
Age Continuous [Mean (Standard Deviation); unit: years] | 17.4 (1.8) | 18.1 (1.9) | 17.8 (1.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 11
  Male | 10 | 10 | 20
Region of Enrollment [Number; unit: participants]
  United States | 15 | 16 | 31
Lean body mass [Mean (Standard Deviation); unit: kg] | 44.03 (11.09) | 44.38 (12.98) | 44.21 (11.90)
Limb fat [Mean (Standard Deviation); unit: kg] | 11.47 (5.49) | 12.92 (9.28) | 12.22 (7.59)
Total body fat [Mean (Standard Deviation); unit: kg] | 24.02 (10.81) | 25.11 (18.29) | 24.58 (14.90)
Trunk fat [Mean (Standard Deviation); unit: kg] | 11.73 (5.58) | 11.40 (9.09) | 11.56 (7.47)
Trunk to limb fat ratio [Mean (Standard Deviation); unit: ratio] | 1.05 (0.29) | 0.87 (0.17) | 0.96 (0.25)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline to Week 24 in Trunk Fat
Time Frame: Baseline to Week 24
Population: Intention To Treat, Last Observation Carried Forward
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Standard Dose Group | High Dose Group
Number analyzed (Participants) | 13 | 15
percent change | -6.27 (12.72) | -8.36 (17.69)
Statistical Analysis 1: Comparison: Standard Dose Group; The null hypothesis (% change in trunk fat (kg) from baseline to Wk24 within the treatment group = 0) was tested against the alternative hypothesis (% change in trunk fat (kg) from baseline to Wk24 within the treatment group ≠0). P-Values for testing this hypothesis for each treatment group are from an analysis of variance (ANOVA) model on ranked data with effects for treatment group, gender and their interaction; Test type: Superiority or Other; p = 0.177, ANOVA
Statistical Analysis 2: Comparison: High Dose Group; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.004, ANOVA

2. Secondary Outcome: Percent Change From Baseline to Week 24 in Lean Body Mass
Time Frame: Baseline to Week 24
Population: Intention To Treat, Last Observation Carried Forward
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Standard Dose Group | High Dose Group
Number analyzed (Participants) | 13 | 15
percent change | 3.85 (4.05) | 7.10 (5.02)
Statistical Analysis 1: Comparison: Standard Dose Group; The null hypothesis (% change in lean body mass (kg) from baseline to Wk24 within the treatment group = 0) was tested against the alternative hypothesis (% change in lean body mass (kg) from baseline to Wk24 within the treatment group ≠0). P-Values for testing this hypothesis for each treatment group are from an analysis of variance (ANOVA) model on ranked data with effects for treatment group, gender and their interaction; Test type: Superiority or Other; p = 0.004, ANOVA
Statistical Analysis 2: Comparison: High Dose Group; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, ANOVA

3. Secondary Outcome: Percent Change From Baseline to Week 24 in Total Body Fat
Time Frame: Baseline to Week 24
Population: Intention To Treat, Last Observation Carried Forward
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Standard Dose Group | High Dose Group
Number analyzed (Participants) | 13 | 15
percent change | -4.62 (9.96) | -9.69 (10.54)
Statistical Analysis 1: Comparison: Standard Dose Group; The null hypothesis (% change in total body fat (kg) from baseline to Wk24 within the treatment group = 0) was tested against the alternative hypothesis (% change in total body fat (kg) from baseline to Wk24 within the treatment group ≠0). P-Values for testing this hypothesis for each treatment group are from an analysis of variance (ANOVA) model on ranked data with effects for treatment group, gender and their interaction; Test type: Superiority or Other; p = 0.653, ANOVA
Statistical Analysis 2: Comparison: High Dose Group; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.002, ANOVA

4. Secondary Outcome: Percent Change From Baseline to Week 24 in Limb Fat
Time Frame: Baseline to Week 24
Population: Intention To Treat, Last Observation Carried Forward
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Standard Dose Group | High Dose Group
Number analyzed (Participants) | 13 | 15
percent change | -3.77 (8.85) | -11.09 (8.97)
Statistical Analysis 1: Comparison: Standard Dose Group; The null hypothesis (% change in limb fat (kg) from baseline to Wk24 within the treatment group = 0) was tested against the alternative hypothesis (% change in limb fat (kg) from baseline to Wk24 within the treatment group ≠0). P-Values for testing this hypothesis for each treatment group are from an analysis of variance (ANOVA) model on ranked data with effects for treatment group, gender and their interaction; Test type: Superiority or Other; p = 0.755, ANOVA
Statistical Analysis 2: Comparison: High Dose Group; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.001, ANOVA

5. Secondary Outcome: Percent Change From Baseline to Week 24 in Trunk to Limb Fat Ratio
Time Frame: Baseline to Week 24
Population: Intention To Treat, Last Observation Carried Forward
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Standard Dose Group | High Dose Group
Number analyzed (Participants) | 13 | 15
percent change | -2.86 (6.77) | 2.92 (16.16)
Statistical Analysis 1: Comparison: Standard Dose Group; The null hypothesis (% change in trunk to limb fat ratio from baseline to Wk24 within the treatment group = 0) was tested against the alternative hypothesis (% change in trunk to limb fat ratio from baseline to Wk24 within the treatment group ≠0). P-Values for testing this hypothesis for each treatment group are from an analysis of variance (ANOVA) model on ranked data with effects for treatment group, gender and their interaction; Test type: Superiority or Other; p = 0.041, ANOVA
Statistical Analysis 2: Comparison: High Dose Group; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.044, ANOVA

ADVERSE EVENTS:
Time Frame: Baseline to Week 28(+/-5 days)
Description: AEs are any untoward medical occurrence in the form of signs, symptoms, abnormal labs or diseases that emerged or worsened relative to baseline (present at the initial study visit) regardless of causal relationship, even if no investigational product was administered. The only SAE occurred approximately 1 month prior to start of study drug.
Arm/Group | Standard Dose Group | High Dose Group
Serious Adverse Events (participants affected / at risk) | 0/15 | 1/16
Other Adverse Events (participants affected / at risk) | 13/15 | 14/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Dose Group (N=15) | High Dose Group (N=16)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Dose Group (N=15) | High Dose Group (N=16)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (2)
Abdominal pain upper (Gastrointestinal disorders) | 1 (2) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dental caries (Infections and infestations) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 1 (1)
Diabetes insipidus (Endocrine disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 2 (3) | 1 (2)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1)
Gynaecomastia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 6 (9) | 6 (11)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Incision site complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Injection site bruising (General disorders) | 2 (2) | 1 (1)
Injection site haemorrhage (General disorders) | 1 (2) | 1 (1)
Insulin resistance (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Insulin-like growth factor increased (Investigations) | 0 (0) | 1 (1)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 3 (4)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 1 (2)
Otitis media (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sinus Headache (Nervous system disorders) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 3 (3)
Tension headache (Nervous system disorders) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 3 (4)
Vaginal infection (Infections and infestations) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days